CLINICAL TRIAL: NCT00220831
Title: Prevention of Diabetic Cardiovascular Complications With Vitamin E 400 IU Treatment to High Risk Patients by Haptoglobin Phenotype (I CARE - Israel Cardiovascular Atherosclerosis Risk and Vitamin E)
Brief Title: Prevention of Cardiovascular Complications in Diabetic Patients With Vitamin E Treatment
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: interim analysis showed significant differences between two treatment groups
Sponsor: Technion, Israel Institute of Technology (Other)
Collaborators: Clalit Health Services (Other); The Kennedy Leigh Charitable Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KL-2004
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes; Myocardial Infarction; Cardiovascular Disease
Keywords: Diabetes; MI; CVD disease
MeSH Terms: conditions — Diabetes Mellitus; Myocardial Infarction; Cardiovascular Diseases

INTERVENTIONS:
Drug: Natural source Vitamin E 400IU/day

SUMMARY:
The purpose of this study is to determine whether Vitamin E treatment to Diabetic patients, who carry the Haptoglobin 2-2 Phenotype, prevents cardiovascular complications such as acute MI and Stroke.

DETAILED DESCRIPTION:
Haptoglobin is a free Hemoglobin scavenger protein. Hemoglobin is an oxidant due to the Fe it carries by the Fenton reaction. Thus it is believed that Haptoglobin is an antioxidant, especially in the site of vascular injury.

Haptoglobin has three phenotype easily identified by a method of gel electrophoresis.

The three phenotype denote as 1-1, 2-1 and 2-2. We have found in several in vitro studies in our lab that Haptoglobin 1-1 is a superior antioxidant over 2-2.

In several large retrospective studies we found that Diabetic patients who are Haptoglobin typed 2-2 have a 5 time risk of having cardiovascular complications (acute MI, CVA, CVD death) over the ones who are Haptoglobin 1-1.

2-1 patients are probably at intermediate risk. While retrospectively typing consecutive serums from patients who participate the HOPE study we found that taking Vitamin E decreased by 50% the CVD incidences of Diabetic patients with the Haptoglobin 2-2 phenotype.

Based on these findings we wish to perform the I CARE study. 5000 diabetic patients aged 55 and above, will be tested for Haptoglobin phenotype.

Knowing the distribution of the different Haptoglobin phenotypes in the Israeli population we estimate that about 2000 will be of the phenotype 2-2.

These 2000 patients will be enrolled in a prospective, doubled blind, randomized and placebo controlled clinical study and will be randomly divided into 2 groups, one receiving Vitamin E 400IU per day and the other receiving matching placebo.

All patients will be followed routinely by their primary physicians in Clalit HMO (the biggest HMO in Israel) in a routine diabetes follow up and treatment (HbA1c, blood pressure control, Lipids, renal function, eye exam for retinopathy etc…) The study steering committee will get anamnestic data and routine tests results every 3 months.

Primary Outcomes: a combination of CVD mortality and non fatal MI and Stroke. Secondary Outcomes: Cardiac Interventions (Angioplasty, Bypass surgery etc…), all cause mortality, heart failure.

Exclusion criteria: 1) patient who takes antioxidant treatment will be asked to stop, or can't be included in the study.

2) Patients who had a CVD incident (MI, Stroke, TIA), Unstable angina pectoris, Uncontrolled HTN, will have to wait a month after stabilization to be included in the study.

3) Allergy to Vitamin E. Follow up duration - 4.5 years. 5% percent of all vitamin receivers will be tested at base line and a year after enrollment, for Vitamin E plasma concentration.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients aged 55 and above

Exclusion Criteria:

* Patient who takes antioxidant treatment will be asked to stop, or can't be included in the study
* Patients who had a CVD incident (MI, Stroke, TIA), Unstable angina pectoris, Uncontrolled HTN, will have to wait a month after stabilization to be included in the study
* Allergy to Vitamin E

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2005-04; Study Completion 2009-12

PRIMARY OUTCOMES:
A combination of CVD mortality non fatal MI and Stoke at a 4 year follow up.

SECONDARY OUTCOMES:
Cardiac Interventions (Angioplasty, Bypass surgery
etc…), all cause mortality, heart failure, at a 4 year follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Uzi Milman, MD, Principal Investigator — Clalit Health Services; Chen Shapira, MD, Study Chair — Clalit Health Services; Shany Blum, MD MSc, Study Chair — Laboratory of Vascular Medicine, the Bruce Rappaport Faculty of Medicine, Technion - Israel Institute of Technology.; Andrew P Levy, MD PhD, Study Chair — Laboratory of Vascular Medicine, the Bruce Rappaport Faculty of Medicine, Technion - Israel Institute of Technology.
Locations (1):
- Clalit Health Services, Haifa and West Galilee - primary health care clinics, in the north of Israel And the Bruce Rappaport Faculty of Medicine, Technion, Haifa, Israel., Haifa, Israel

REFERENCES:
- [Background] Melamed-Frank M, Lache O, Enav BI, Szafranek T, Levy NS, Ricklis RM, Levy AP. Structure-function analysis of the antioxidant properties of haptoglobin. Blood. 2001 Dec 15;98(13):3693-8. doi: 10.1182/blood.v98.13.3693. PMID 11739174
- [Background] Levy AP, Roguin A, Hochberg I, Herer P, Marsh S, Nakhoul FM, Skorecki K. Haptoglobin phenotype and vascular complications in patients with diabetes. N Engl J Med. 2000 Sep 28;343(13):969-70. doi: 10.1056/NEJM200009283431313. No abstract available. PMID 11012324
- [Background] Nakhoul FM, Marsh S, Hochberg I, Leibu R, Miller BP, Levy AP. Haptoglobin genotype as a risk factor for diabetic retinopathy. JAMA. 2000 Sep 13;284(10):1244-5. doi: 10.1001/jama.284.10.1244-a. No abstract available. PMID 10979109
- [Background] Nakhoul FM, Zoabi R, Kanter Y, Zoabi M, Skorecki K, Hochberg I, Leibu R, Miller B, Levy AP. Haptoglobin phenotype and diabetic nephropathy. Diabetologia. 2001 May;44(5):602-4. doi: 10.1007/s001250051666. PMID 11380078
- [Background] Roguin A, Hochberg I, Nikolsky E, Markiewicz W, Meisel SR, Hir J, Grenadier E, Beyar R, Levy AP. Haptoglobin phenotype as a predictor of restenosis after percutaneous transluminal coronary angioplasty. Am J Cardiol. 2001 Feb 1;87(3):330-2, A9. doi: 10.1016/s0002-9149(00)01368-0. PMID 11165970
- [Background] Levy AP, Hochberg I, Jablonski K, Resnick HE, Lee ET, Best L, Howard BV; Strong Heart Study. Haptoglobin phenotype is an independent risk factor for cardiovascular disease in individuals with diabetes: The Strong Heart Study. J Am Coll Cardiol. 2002 Dec 4;40(11):1984-90. doi: 10.1016/s0735-1097(02)02534-2. PMID 12475459
- [Background] Hochberg I, Roguin A, Nikolsky E, Chanderashekhar PV, Cohen S, Levy AP. Haptoglobin phenotype and coronary artery collaterals in diabetic patients. Atherosclerosis. 2002 Apr;161(2):441-6. doi: 10.1016/s0021-9150(01)00657-8. PMID 11888529
- [Background] Levy AP, Gerstein HC, Miller-Lotan R, Ratner R, McQueen M, Lonn E, Pogue J. The effect of vitamin E supplementation on cardiovascular risk in diabetic individuals with different haptoglobin phenotypes. Diabetes Care. 2004 Nov;27(11):2767. doi: 10.2337/diacare.27.11.2767. No abstract available. PMID 15505023
- [Derived] Milman U, Blum S, Shapira C, Aronson D, Miller-Lotan R, Anbinder Y, Alshiek J, Bennett L, Kostenko M, Landau M, Keidar S, Levy Y, Khemlin A, Radan A, Levy AP. Vitamin E supplementation reduces cardiovascular events in a subgroup of middle-aged individuals with both type 2 diabetes mellitus and the haptoglobin 2-2 genotype: a prospective double-blinded clinical trial. Arterioscler Thromb Vasc Biol. 2008 Feb;28(2):341-7. doi: 10.1161/ATVBAHA.107.153965. Epub 2007 Nov 21. PMID 18032779